CLINICAL TRIAL: NCT02473406
Title: Thymosin Alpha 1 in the Prevention of Pancreatic Infection Following Acute Necrotizing Pancreatitis
Acronym: TRACE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weiqin Li (Other)
Collaborators: The First Affiliated Hospital of Nanchang University (Other); The Affiliated Hospital of Qingdao University (Other); Zunyi Medical College (Other); the Affiliated Nanhua Hospital, University of South China (Unknown); Second Affiliated Hospital of Nantong University (Other); Wannan Medical College Yijishan Hospital (Other); the 908th Hospital of Chinese People's Liberation Army Joint Logistic Support Force (Unknown); Jiangsu Province Hospital of Traditional Chinese Medicine (Other); Zhejiang Provincial People's Hospital (Other); Luoyang Central Hospital (Other); The Affiliated Hospital of Henan University of Science and Technology (Unknown); Clinical Medical College of Yangzhou University (Unknown); The First People's Hospital of Shangqiu (Unknown); Qilu Hospital of Shandong University (Other); The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Sponsor-Investigator, Weiqin Li, Professor, Nanjing University School of Medicine
Organization: Nanjing University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TRACE trial
Record Dates: First submitted 2015-06-12; First posted 2015-06-16 (Estimated); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Pancreatitis, Acute Necrotizing
Keywords: Acute Pancreatitis, prevent,Necrotizing
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing; Pancreatitis | interventions — Thymalfasin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thymosin (Experimental): Thymosin alpha 1 has been shown to have immunomodulatory properties
  Interventions: Drug: Thymosin Alpha 1
- Placebo (Placebo Comparator): normal saline;
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Thymosin Alpha 1 — In addition to the standard treatment, thymosin therapy will be started after admission: 1.6mg I.H q12h for the first 7 days and 1.6mg I.H, qd for the following 7 days or until discharge.
  Other Names: Thymosin Group
  Arms: Thymosin
Drug: normal saline — Placebo inject will be given at the same dose as Thymosin in addition to the standard treatment.
  Other Names: Placebo Group
  Arms: Placebo

SUMMARY:
Infected pancreatic necrosis and its related septic complications are the major cause of death in patients with acute pancreatitis, therefore prevention of pancreatic infection is of great clinical value in the treatment of AP.

Immunosuppression and disorders characterized by decreased HLA-DR expression and unbalanced CD3/CD4+/CD8+ T cells of PBMC are thought to be associated with the development of pancreatic infection. Thymosin alpha 1 has been shown to have immunomodulatory properties and its effects in preventing pancreatic infection was not well studied. To evaluate the effects of TA1 use in the early phase on preventing pancreatic infection, immunomodulation and clinical outcomes in patients with AP,we aimed to design this study.

DETAILED DESCRIPTION:
Study Background & Rationale:

Infected pancreatic necrosis and its related septic complications are the major cause of death in patients with acute pancreatitis1, therefore prevention of pancreatic infection is of great clinical value in the treatment of AP.

Immunosuppression and disorders characterized by decreased HLA-DR expression and unbalanced CD3/CD4+/CD8+ T cells of PBMC are thought to be associated with the development of pancreatic infection2, 3. Thymosin alpha 1 has been shown to have immunomodulatory properties and its effects in preventing pancreatic infection was not well studied4.

Aim of This Study:

To evaluate the effects of TA1 use in the early phase on preventing pancreatic infection, immunomodulation and clinical outcomes in patients with AP.

Sample Size Estimation:

The prevalence of pancreatic infection was reported to be around 25% in AP episodes. To demonstrate a 40% reduction in the prevalence of pancreatic infection with 80% power at a two-sided alpha level of .05, we projected an estimated sample size of 500 participants. Considering possible 2% withdraw, we plan to randomize 510 patients in total.

ELIGIBILITY:
Inclusion criteria

1. Symptoms and signs of acute pancreatitis based on abdominal pain suggestive of AP, serum amylase at least three times the upper limit of normal, and/or characteristic findings of AP on computed tomography or less commonly magnetic resonance imaging (MRI) or transabdominal ultrasonography according to the Revised Atlanta Criteria[15];
2. Less than one week from the onset of abdominal pain;
3. Age between 18 to 70 years old;
4. Acute Physiology and Chronic Health Evaluation(APACHE II) score ≥8 during the last 24 hours before enrollment
5. Balthazar CT score ≥5 (presence of pancreatic necrosis)[16].
6. Written informed consent obtained

Exclusion criteria

1. Pregnant pancreatitis;
2. History of chronic pancreatitis；
3. Malignancy related acute pancreatitis
4. Receiving early intervention or surgery due to abdominal compartment syndrome or other reasons before admission；
5. Patients with a known history of severe cardiovascular, respiratory, renal or hepatic diseases defined as (1) greater than New York Heart Association Class II heart failure(Class II not included), (2) active myocardial ischemia or (3) cardiovascular intervention within previous 60 days, (4) history of cirrhosis or (5) chronic kidney disease with creatinine clearance< 40 mL/min, or (6) chronic obstructive pulmonary disease with requirement for home oxygen;
6. Patients with preexisting immune disorders such as AIDS.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2020-12-24 (Actual); Study Completion 2021-03-24 (Actual)

PRIMARY OUTCOMES:
Occurrence of pancreatic infection: | during the index admission

SECONDARY OUTCOMES:
The occurrence of new-onset organ failure and new-onset persistent organ failure | during the index admission
  (SOFA score for respiration, cardiovascular, or renal system ≥2 ). New-onset is defined as events that occur after randomization and not present 24 hours before randomization
In-hospital mortality | during the index admission
Bleeding requiring intervention | during the index admission
Gastrointestinal perforation or fistula requiring intervention | during the index admission
Incidence of pancreatic fistula | during the index admission
New receipt of mechanical ventilation/renal replacement therapy /New receipt of vasoactive agents | during the index admission
  not applied 24 hours before randomization
The requirement for catheter drainage/Number of drainage procedures required | during the index admission
The requirement for minimally-invasive debridement/Number of minimally invasive necrosectomy required | during the index admission
The requirement for open surgery/Number of open surgery required | during the index admission
Length of intensive care unit(ICU) stay/Length of hospital stay | during the index admission
SOFA score/ CRP level/ HLA-DR level/ Lymphocyte count | on day0, day7, and day14
In-hospital cost. | during the index admission
Incidence of infection within 90 days after enrollment | 90 days after enrollment
Mortality within 90 days after enrollment | 90 days after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Li Weiqin, M.D., Study Chair — Department of SICU, Research Institute of General Surgery Jinling Hospital, Nanjing, Jiangsu, Chin; Ke Lu, M.D., Study Director — Department of SICU, Research Institute of General Surgery Jinling Hospital, Nanjing, Jiangsu, Chin; Zhou Jing, M.D., Principal Investigator — Department of SICU, Research Institute of General Surgery Jinling Hospital, Nanjing, Jiangsu, Chin
Locations (2):
- China (2):
  - Department of SICU, Research Institute of General Surgery Jinling Hospital, Nanjing, Jiangsu, China, Nanjing, Jiangsu
  - Jinling Hospital, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Huang X, Mao W, Hu X, Qin F, Zhao H, Zhang A, Wang X, Stoppe C, Zhou D, Ke L, Ni H; Chinese Acute Pancreatitis Clinical Trials Group (CAPCTG). Immune-Enhancing Treatment among Acute Necrotizing Pancreatitis Patients with Metabolic Abnormalities: A Post Hoc Analysis of a Randomized Clinical Trial. Gut Liver. 2024 Sep 15;18(5):906-914. doi: 10.5009/gnl230326. Epub 2024 Feb 15. PMID 38356344
- [Derived] Ke L, Mao W, Shao F, Zhou J, Xu M, Chen T, Liu Y, Tong Z, Windsor J, Ma P, Li W; Chinese Acute Pancreatitis Clinical Trials Group (CAPCTG). Association between pretreatment lymphocyte count and efficacy of immune-enhancing therapy in acute necrotising pancreatitis: a post-hoc analysis of the multicentre, randomised, placebo-controlled TRACE trial. EClinicalMedicine. 2023 Mar 24;58:101915. doi: 10.1016/j.eclinm.2023.101915. eCollection 2023 Apr. PMID 37007743
- [Derived] Zhou J, Mao W, Ke L, Chen T, He W, Pan X, Chen M, He C, Gu W, Wu J, Song J, Ni H, Tu J, Sun J, Zhang G, Chen W, Xue B, Zhao X, Shao M, Liu Y, Tong Z, Li W; Chinese Acute Pancreatitis Clinical Trials Group (CAPCTG). Thymosin alpha 1 in the prevention of infected pancreatic necrosis following acute necrotising pancreatitis (TRACE trial): protocol of a multicentre, randomised, double-blind, placebo-controlled, parallel-group trial. BMJ Open. 2020 Sep 29;10(9):e037231. doi: 10.1136/bmjopen-2020-037231. PMID 32994239